CLINICAL TRIAL: NCT01227551
Title: A Phase 2 Study of the Efficacy and Safety of Intratumoral CAVATAK™ (Coxsackievirus A21, CVA21) in Patients With Stage IIIc and Stage IV Malignant Melanoma (VLA-007 CALM )
Brief Title: A Study of Intratumoral CAVATAK™ in Patients With Stage IIIc and Stage IV Malignant Melanoma (VLA-007 CALM )
Acronym: CALM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Viralytics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: V937-006; VLA-007 (Other: Viralytics Study ID)
Record Dates: First submitted 2010-10-20; First posted 2010-10-25 (Estimated); Results first posted 2017-05-15 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-06

CONDITIONS: Malignant Melanoma
Keywords: Melanoma; CALM
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intratumoral injection (Experimental): Each patient will receive 4 separate Coxsackievirus A21 (CVA21) administrations in the first 8 days on trial (Days 1, 3, 5 and 8), followed by a fifth dose 2 weeks later (Day 22) and further administrations at 3 weekly intervals (Days 43, 64, 85, 106 and 127, up to a maximum of 10 sets of injections) until confirmed disease progression or development of excessive toxicity. Subjects with stable disease or better at Day 127 were eligible to receive up 9 more sets of CVA21 administrations under an extension protocol (VLA-008).
  Interventions: Biological: Coxsackievirus A21 (CVA21)

INTERVENTIONS:
Biological: Coxsackievirus A21 (CVA21) — CVA21 is a live oncolytic virus preparation derived from the non-genetically altered prototype Kuykendall strain of Coxsackievirus A21.

SUMMARY:
The purpose of this study is to assess the clinical efficacy of Intratumoral (IT) CVA21 in terms of immune-related Progression-Free Survival (irPFS) at 6 months as monitored via immune-related Response Criteria [irRECIST 1.1] (revised Response Evaluation Criteria In Solid Tumors [RECIST] 1.1).

DETAILED DESCRIPTION:
This is a multicenter, open-label, 2-stage, single-arm efficacy and safety study. Approximately 63 patients with histologically proven stage IIIc or stage IV melanoma who fail to qualify for curative surgery and who bear one or more tumors that are accessible for direct injections and at least one measurable lesion by RECIST 1.1 criteria will be considered.

Prospective patients will attend the study center for initial screening within 28 days prior to treatment with CVA21. They will have the nature of the study and its procedures and risks fully explained. All patients must provide a written informed consent to participate in the study.

The dose of CVA21 for this study is 3 x 108 TCID50 (about 4.5 x 106 TCID50/kg for a 70-kg patient) by IT administration. Each patient will receive 4 separate CVA21 administrations in the first 8 days on trial (Days 1, 3, 5 and 8), followed by a fifth dose 2 weeks later (Day 22) and further administrations at 3 weekly intervals (Days 43, 64, 85, 106 and 127, up to a maximum of 10 sets of injections) or until confirmed disease progression or development of excessive toxicity.

Disease status will be assessed by contrast-enhanced computerized tomography (CT) or magnetic resonance imaging (MRI) scan and/or direct caliper measurement (and ultrasound assistance, if necessary) and categorized by immune-related RECIST 1.1 criteria prior to commencing treatment (baseline) and at Days 43, 85, 127 and 169 and 12-weekly intervals thereafter until disease progression. At 2 years, intervals can increase to 6 months.

At 12 weeks post-commencement of treatment (Day 85), if a patient's disease status is classed as progressive disease (but without rapid clinical deterioration) the patient may remain on the trial for a further 6 weeks, when his/her disease status will be confirmed prior to the scheduled treatment. If disease progression is confirmed, the patient will cease treatment but will remain on the study and be observed for efficacy and safety until initiation of treatment with non-CVA21 anticancer therapies. However, survival will be followed until death. If stable disease or better (CR or PR) is observed at this time, the patient will continue treatment as per the protocol. Complete and partial responses will be confirmed at the next contrast-enhanced CT or MRI scan analysis.

Patients who have evidence of biologic activity, i.e., tumor inflammatory reaction and/or stable disease or better, at 18 weeks (Day 127) are eligible to participate in the extension trial in which they will continue to receive IT injections of CVA21 every 3 weeks up to a total of 1 year of therapy from the first injection.

Throughout the trial, immunological responses to the tumor and CVA21 will be monitored.

After the full CVA21 injection schedule has been completed, patients will be followed at 12-weekly intervals beginning on Day 169 for a total of 12 months according to the schedule for safety assessment and indefinitely for survival. Patients with progressive disease (but without rapid clinical deterioration) at 6 months (Day 169) will have a further tumor assessment 6 weeks later for confirmation or continuation of observation for duration of disease control and all subjects will be followed for survival. Patients who are withdrawn from treatment with CVA21 during the treatment phase must also be followed up every 6 weeks for 12 weeks for safety and for survival.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with histologically proven stage IIIc or stage IV melanoma who fails to qualify for curative surgery and who bears one or more tumors that are accessible for direct injection
2. Patient must have had no more than one previous systemic regimen for management of melanoma; however, adjuvant chemotherapy administered 6 months or longer before entering the trial does not count as a line of treatment
3. Absence of circulating serum neutralizing antibodies to CVA21 (titer < 1:16)
4. At least one tumor 0.5 to 10 cm in the longest diameter must be suitable for injection and at least one tumor must be equal to or greater than 1 cm and qualified to be a target lesion for RECIST 1.1 criteria
5. Patient must have adequate hematologic, hepatic and renal function, defined as:

   * Absolute neutrophil count (ANC) > 1.5 x 10^9/L, platelets > 100 x 10^9/L
   * Bilirubin < 1.5 times the upper limit of normal (ULN), aspartate aminotransferase (AST) < 2.5 x ULN
   * Serum creatinine < 1.5 x ULN; if > 1.5 x ULN, it must be confirmed that creatinine clearance > 30 mL/minute
6. Serum lactate dehydrogenase (LDH) levels < or = 1.5 x ULN
7. Male or female age 18 years or older
8. Performance status (Eastern Cooperative Oncology Group [ECOG]) 0 or 1
9. Estimated life expectancy of more than 6 months
10. Recovered from prior therapy with at least 4 weeks since the last exposure to chemotherapy or radiotherapy
11. Patient is able and willing to provide written informed consent to participate in the study
12. Fertile males and females must agree to the use of an adequate form of contraception, e.g., condoms for males. A negative pregnancy test is required in female patients of childbearing potential.

Exclusion Criteria:

1. Mucosal or ocular primary tumors
2. Bone metastases
3. Greater than 3 visceral metastases
4. Any visceral metastases > 10 cm
5. Serum anti-CVA21 neutralizing titer of > 1:16 at baseline
6. Presence of any central nervous system (CNS) tumor that has not been stable for at least 3 months off corticosteroids and confirmed by imaging
7. Tumors to be injected lying in mucosal regions or close to an airway, major blood vessel or spinal cord that, in the opinion of the Investigators, could cause occlusion into a major vessel in the case of necrosis
8. Only measurable tumor had prior local radiotherapy without subsequent nodule progression
9. Patient has received chemotherapy within the last 4 weeks prior to first injection
10. ECOG score greater than 1
11. Estimated life expectancy of less than 6 months
12. Pregnancy or breastfeeding
13. Primary or secondary immunodeficiency, including immunosuppressive disease, and immunosuppressive doses of corticosteroids (e.g., prednisolone > 7.5 mg per day) or other immunosuppressive medications including cyclosporine, azathioprine, interferons within the past 4 weeks prior to screening
14. Positive serology for human immunodeficiency virus (HIV), hepatitis B or C
15. Full dose anticoagulation or a history of bleeding diathesis or poorly controlled bleeding in the last month prior to screening
16. Previous splenectomy
17. Presence of uncontrolled infection
18. Presence of unstable neurological disease
19. Any uncontrolled medical condition that, in the opinion of the investigator, is likely to place the patient at unacceptable risk during the study or reduce his/her ability to complete the study
20. Participation in another study requiring administration of an investigational drug or biological agent within the last 4 weeks prior to screening
21. Any other medical or psychological condition that would preclude participation in the study or compromise ability to give informed consent
22. Participation in any previous melanoma immunotherapy trial within 1 month prior to entry to this trial or any trial of any other investigational agent within the last month prior to entry to this trial
23. Active infections or serious general medical conditions
24. Patients with previous malignancies should only be permitted if they have been in a continued state of "no evidence of disease" for at least 5 years with the exception of adequately treated carcinoma in situ of the cervix, ductal carcinoma in situ (DCIS) of the breast, and basal cell/squamous cell skin cancer
25. Known allergy to treatment medication or its excipients and/or to the contrast medium

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2011-12-29 (Actual); Primary Completion 2016-04-06 (Actual); Study Completion 2016-04-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Andtbacka, MD, Principal Investigator — Associate Professor
Locations (10):
- United States (10):
  - Moores UCSD Cancer Center, La Jolla, California
  - St Mary's Medical Center, San Francisco, California
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Oncology Specialists, SC, Niles, Illinois
  - Investigative Clinical Research of Indiana, Indianapolis, Indiana
  - Atlantic Melanoma Center, Morristown, New Jersey
  - Providence Cancer Center, Portland, Oregon
  - Mary Crowley Cancer Research Centers, Dallas, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Andtbacka RHI, Curti B, Daniels GA, Hallmeyer S, Whitman ED, Lutzky J, Spitler LE, Zhou K, Bommareddy PK, Grose M, Wang M, Wu C, Kaufman HL. Clinical Responses of Oncolytic Coxsackievirus A21 (V937) in Patients With Unresectable Melanoma. J Clin Oncol. 2021 Dec 1;39(34):3829-3838. doi: 10.1200/JCO.20.03246. Epub 2021 Aug 31. PMID 34464163

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from medical clinics from 27-Dec-2011 to 29-Jul-2015 (last subject enrolled in VLA-008).
Pre-assignment Details: Subjects were screened for and excluded from the study if they had pre-existing antibodies to CVA21.
Groups:
- CVA21: CVA21 monotherapy
Period: Overall Study
Arm/Group | CVA21
Started | 57
Completed | 23
Not Completed | 34

BASELINE CHARACTERISTICS:
Arm/Group | CVA21
Number analyzed (Participants) | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.7 (14.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 56
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 56
  More than one race | 0
  Unknown or Not Reported | 0
Height [Mean (Standard Deviation); unit: centimeters] | 172.7 (11.84)
Weight [Mean (Standard Deviation); unit: kilograms] | 86.16 (21.869)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Immune-related Progression-Free Survival (irPFS) at 6 Months
Description: To assess the clinical efficacy of Intratumoral (IT) CVA21 in terms of immune-related Progression-Free Survival (irPFS) at 6 months.
Time Frame: 6 months
Population: ITT Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CVA21
Number analyzed (Participants) | 57
percentage of participants | 38.6 [26.0 to 52.4]

2. Secondary Outcome: Durable Response Rate
Description: Per Immune-Related Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT/MRI or calipers: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Durable Response Rate (DRR) = CR + PR.
Time Frame: 6 months or more
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | CVA21
Number analyzed (Participants) | 57
percentage of participants | 21.1

ADVERSE EVENTS:
Time Frame: 1 year
Description: Listed SAEs and AEs are irrespective of treatment relationship. No SAEs reported were attributable to CVA21. No SUSARs were reported for the VLA-007/008 study.
Arm/Group | CVA21
Serious Adverse Events (participants affected / at risk) | 11/57
Other Adverse Events (participants affected / at risk) | 54/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CVA21 (N=57)
squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
cardiac arrest (Cardiac disorders) | 1 (1)
cardiogenic shock (Cardiac disorders) | 1 (1)
abdominal pain (Gastrointestinal disorders) | 1 (1)
nausea (Gastrointestinal disorders) | 1 (1)
vomiting (Gastrointestinal disorders) | 1 (1)
fatigue (General disorders) | 1 (1)
bacteremia (Infections and infestations) | 1 (1)
cellulitis (Infections and infestations) | 1 (1)
sepsis (Infections and infestations) | 1 (1)
metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
haemorrhage intracranial (Nervous system disorders) | 1 (1)
motor dysfunction (Nervous system disorders) | 1 (1)
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CVA21 (N=57)
anaemia (Blood and lymphatic system disorders) | 5 (7)
iron deficiency (Blood and lymphatic system disorders) | 4 (4)
constipation (Gastrointestinal disorders) | 7 (7)
diarrhoea (Gastrointestinal disorders) | 8 (8)
nausea (Gastrointestinal disorders) | 8 (11)
vomiting (Gastrointestinal disorders) | 7 (8)
chills (General disorders) | 16 (27)
fatigue (Gastrointestinal disorders) | 23 (33)
influenza like illness (General disorders) | 5 (7)
injection site discharge (General disorders) | 3 (4)
injection site erythema (General disorders) | 8 (11)
injection site oedema (General disorders) | 3 (4)
injection site pain (General disorders) | 18 (49)
injection site pruritus (General disorders) | 3 (7)
injection site reaction (General disorders) | 3 (3)
malaise (General disorders) | 4 (4)
oedema peripheral (General disorders) | 3 (3)
pain (General disorders) | 11 (13)
pyrexia (General disorders) | 7 (7)
rhinitis (Infections and infestations) | 3 (3)
upper respiratory tract infection (Infections and infestations) | 5 (6)
decreased appetite (Metabolism and nutrition disorders) | 6 (8)
arthralgia (Musculoskeletal and connective tissue disorders) | 6 (7)
back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
myalgia (Musculoskeletal and connective tissue disorders) | 9 (11)
neck pain (Musculoskeletal and connective tissue disorders) | 3 (4)
pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (5)
dizziness (Nervous system disorders) | 9 (10)
headache (Nervous system disorders) | 12 (16)
anxiety (Psychiatric disorders) | 4 (4)
cough (Respiratory, thoracic and mediastinal disorders) | 6 (8)
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 (8)
sinus congestion (Respiratory, thoracic and mediastinal disorders) | 4 (4)
hyperhidrosis (Skin and subcutaneous tissue disorders) | 5 (8)
pruritus (Skin and subcutaneous tissue disorders) | 6 (7)
rash (Skin and subcutaneous tissue disorders) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other